CLINICAL TRIAL: NCT03966573
Title: Femoral Lengthening Might Impair Physical Function and Lead to Structural Changes in Adjacent Joints; 10 Patients With 27 to 34 Years Follow-up.
Brief Title: Femoral Lengthening Might Impair Physical Function and Lead to Structural Changes in Adjacent Joints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sophies Minde Ortopedi (Industry)
Responsible Party: Principal Investigator, Patrick Aleksander Bjørge, Physiotherapist, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018/416
Record Dates: First submitted 2019-03-19; First posted 2019-05-29 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Leg Length Inequality; Leg; Lengthening; Osteoarthritis, Knee; Osteoarthritis of Hip; Quality of Life
MeSH Terms: conditions — Leg Length Inequality; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Phantoms, Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluating function, Radiographic imaging, Forms (Other): * Tests for lower extremity function
  * Evaluating arthritis of hip and knee, leg length discrepancy and axis deviation radiographically
  * Evaluating quality of life, function and pain by forms
  Interventions: Radiation: Radiographic imaging; Other: Evaluating function; Other: Forms

INTERVENTIONS:
Radiation: Radiographic imaging — Evaluating arthritis in knee and hip bilaterally. Evaluating axis deficiancy and leg length discrepancy.
  Other Names: Knee front; knee side; lower extremity axis front; lower extremity axis side; pelvis front
Other: Evaluating function — Test function and physical capasity
  Other Names: 30 seconds sit to stand; single leg hop test; stair test; goniometric ROM measurement hip and knee
Other: Forms — Forms for evaluating quality of life, pain, function
  Other Names: EQ-5D-5L; KOOS - knee osteoarthritis outcome score; IPAQ - international physical activity questionnaire

SUMMARY:
This study evaluates function, quality of life and development of hip- and knee osteoarthritis minimum 15 years after unilateral femoral lengthening on people with idiopathic or post-traumatic anisomelia.

DETAILED DESCRIPTION:
This study has a cross-sectional design, where patients that completed femoral lengthening more than 15 years ago and fulfills the inclusion criteria's are invited to participate. Patients will undergo radiographic imaging to evaluate hip- and knee arthritis, axis deviaton and leg length discrepancy. To evaluate quality of life, function and pain, the participants will complete the forms EQ-5D-5L, Knee osteoarthritis outcome score (KOOS) and International physical activity questionnaire (IPAQ). Bilateral active hip and knee range of motion will be measured with hand held goniometer, and the functional tests 30 seconds sit to stand, hop tests and stair test will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic or post traumatic leg length discrepancy who are lengthened with the callutasis method minimum 15 years ago

Exclusion Criteria:

* Patients that are lenghtened with innate pathology resulting in shortening of the limb, angle deviation and less musculature, for example congenital femoral deficiency or fibula hemimelia.
* Patients with acquired leg length discrepancy who have had infection in knee or hip joint

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
hip or knee osteoarthritis | One day
  Radiographic imaging. Kellgren & Lawrence classification and joint space width will be measured
Lower extremity strength | one day
  30 seconds sit to stand test, measuring strength in lower extremities
Lower extremity function | one day
  Single leg hop tests
Aerob capasity | one day
  Stair test, 18 steps up and down three times
measure of health related quality of life with EQ-5D-5L | one day
  participants report the extent of problems they have with endpoints 1-5, where 1 is no problems and 5 is not able to in the five dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The questionnaire also contains a vertical analogue scale with the labelled endpoints 0-100 where 0 is the worst imaginable health state and 100 the best imaginable health state, giving a valuation of the participants own health state that can be used as a quantitative measure of health outcome based on the patients' own judgement
measure of function and pain with Knee Osteoarthritis Outcome Score (KOOS) | one day
  The participant answer questions regarding pain, function, stiffness and quality of life regarding knee pain. Endpoints 0 - 4, where 0 indicate no problems and 4 indicate extreme problems
measuring physical activity level with International Physical Activity Questionnaire (IPAQ) | one day
  Participants answer the amount of time being in vigorous activity, moderate activity, walking and sitting during the last 7 days. Answers are given in number of days in each of the activity categories, and time in hours and minutes on a regular day the actual week
Active range of motion | one day
  Hand held goniometric measurement of active range of motion in hip and knee bilaterally

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
IDP that underlie results in a publication
Time Frame: Data will become avaliable within 6 months of study completion
Access Criteria: Shared in an open access publication

REFERENCES:
- [Derived] Bjorge PA, Tveter AT, Steen H, Gunderson R, Horn J. Femoral lengthening might impair physical function and lead to structural changes in adjacent joints: 10 patients with 27 to 34 years' follow-up. Acta Orthop. 2021 Jun;92(3):329-334. doi: 10.1080/17453674.2020.1866864. Epub 2021 Jan 7. PMID 33410356

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03966573/Prot_SAP_000.pdf